CLINICAL TRIAL: NCT00178217
Title: Music Therapy as Procedural Support During Botulinum Injections for Pediatric Patients
Brief Title: Music Therapy During Botulinum Injections
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Joan And Harold Feinbloom Supporting Foundation (Other)
Responsible Party: Principal Investigator, OJ Sahler, Professor of Pediatrics, Psychiatry, Medical Humanities & Oncology, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 9507
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Cerebral Palsy
Keywords: Botulinum Toxin; Music Therapy; Cerebral Palsy; Procedural Support
MeSH Terms: conditions — Cerebral Palsy | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy (Experimental): The music therapy intervention will consist of approximately 30 minutes of active music making and/or improvisation. The session will begin at least 15 minutes prior to receiving the Botox injections, followed by the necessary time of the procedure and 10 minutes following. During this time the patient will be encouraged to actively engage in a musical activity of his/her choice. After the last injection has been administered, the monitoring and music therapy will continue for up to 10 minutes, and focus on soothing and relaxation rather than on distraction.
  Interventions: Behavioral: Music Therapy
- Standard Care Control (No Intervention): Subjects will receive standard care at control condition sessions, which includes the use of television, books, CD's, a child life specialist (when available) or other activities to help cope with the procedure.

INTERVENTIONS:
Behavioral: Music Therapy — The music therapy intervention will consist of approximately 30 minutes of active music making and/or improvisation. The session will begin at least 15 minutes prior to receiving the Botox injections, followed by the necessary time of the procedure and 10 minutes following. During this time the patient will be encouraged to actively engage in a musical activity of his/her choice. After the last injection has been administered, the monitoring and music therapy will continue for up to 10 minutes, and focus on soothing and relaxation rather than on distraction.
  Arms: Music Therapy

SUMMARY:
The primary objectives for this study are:

1. To demonstrate that music therapy can be an effective means of procedural support for children undergoing botox injections.
2. To explore patient, parent and healthcare personnel satisfaction with music therapy as procedural support.
3. To assess the influence of music therapy on physiologic (blood pressure, oxygen saturation, heart rate) and emotional (crying time) responses of patients.

DETAILED DESCRIPTION:
Many children with spastic Cerebral Palsy and other types of muscle dystonia are injected with Botulinum toxin A (Botox) to reduce pathological reflexes and improve muscle function. Such treatment requires injections to each affected muscle group, which can be both painful and distressing. Music therapy has been shown to reduce pain and decrease stress and anxiety for pediatric patients undergoing other types of medical procedures.

The goal of this study is to determine whether music therapy can be effectively integrated as a means of procedural support during Botox injections. This study investigates the efficacy of music therapy in reducing manifestations of pain during Botox injections. Secondary benefits may include increased satisfaction among medical personnel and parents.

Patients between the ages of 2-17 being treated with Botox were eligible for enrollment. Prior to the start of this study, patients had the option of receiving music therapy support during their Botox injections; these subjects continued to receive music therapy upon enrolling in the study. Subjects who had not previously received music therapy were videotaped for two Botox sessions before having a music therapy intervention. The percentage of crying time during the procedure was calculated from videotapes taken during the sessions. Surveys were given to parent/guardians and the healthcare provider performing the procedure to provide feedback on the effectiveness of the music intervention for the child and themselves.

Comparing average crying times for 44 children's first study visit with or without music therapy shows that children who receive music therapy cry less than children who do not, although the difference is not statistically significant. Both parent and healthcare provider surveys indicate a high level of satisfaction with the music therapy intervention.

The current data indicate that music therapy may be a highly effective means of procedural support, but strong conclusions cannot be drawn without more data.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for diplegic or hemiplegic cerebral palsy or muscle spasticity resulting from brain injury, with Botulinum toxin injections.

Exclusion Criteria:

* None

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2002-07; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Music therapy will be effectively integrated as a means of procedural support for children undergoing botox injections with a success rate of 80% in enrolling, treating and collecting data from study subjects. | End of study
Music therapy will increase satisfaction by decreasing the distress related to botox injections for child, parent and medical staff. | From beginning to end of session
Subjects receiving music therapy will demonstrate less procedure-related distress as manifested by: Less of an increase in blood pressure and heart rate, less of a decrease in oxygen saturation, and a lower proportion of procedure time spent crying | From beginning to end of session

SECONDARY OUTCOMES:
When patients receive music therapy, they will be more likely to undergo Botox injections without the use of sedation. | By end of study

CONTACTS AND LOCATIONS:
Overall Officials: Olle Jane Z Sahler, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Sahler OJZ, Hunter BC, Oliva R, Du C, Hoffman T, Liptak G, Cole,LL. "Music Therapy as Procedural Support During Botulinum Toxin Injections". Pediatric Academic Societies. Pediatr Res 2004; 55:87A, Abstract 492.
- See also: American Music Therapy Association Home Page — http://www.musictherapy.org/